CLINICAL TRIAL: NCT03093415
Title: A Prospective Cohort Study Comparing the Effectiveness of Zepatier for the Treatment of Hepatitis C in an Academic Center Population to People Who Inject Drugs (PWIDs) in a Safety Net Clinic Setting Engaged in Either a Medication Assisted Therapy (MAT) or Syringe Exchange Program
Brief Title: Hepatitis C Treatment in PWIDs: MAT or Syringe Exchange Assisted-therapy vs Standard of Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Andrew Seaman, Co Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRS00002743
Record Dates: First submitted 2017-03-09; First posted 2017-03-28 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C; Substance Use Disorders; Substance Abuse, Intravenous
Keywords: Hepatitis C; HCV; People Who Inject Drugs; PWID; Medication Assisted Therapy; MAT; Needle Exchange Program
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders; Substance Abuse, Intravenous | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Intervention Model Description: Two parallel investigational groups in different community health clinic treatment settings assigned to treatment with elbasvir-grazoprevir as compared to an academic hepatology clinic retrospective cohort treated with elbasvir-grazoprevir.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Old Town Clinic, Medication Assisted Therapy group (Active Comparator): 25 People Who Inject Drugs engaged in a Medication Assisted Therapy treatment program for their substance use disorder, treated for their HCV using elbasvir-grazoprevir (50 mg/100 mg) for 12 weeks.
  Interventions: Drug: elbasvir-grazoprevir (50 mg/100 mg)
- Outside In Clinic, Needle Exchange Program (Active Comparator): 25 People Who Inject Drugs engaged in a Needle Exchange Program with risk reduction education, treated for their HCV using elbasvir-grazoprevir (50 mg/100 mg) for 12 weeks.
  Interventions: Drug: elbasvir-grazoprevir (50 mg/100 mg)
- OHSU Hepatology Clinic, Academic center Retrospective Cohort (Other): 50 people with substance use disorder and HCV engaged with an Academic Hepatology Clinic (Oregon Health & Sciences University, OHSU) and treated with elbasvir-grazoprevir (50 mg/100 mg) for 12 weeks.
  Interventions: Drug: elbasvir-grazoprevir (50 mg/100 mg)

INTERVENTIONS:
Drug: elbasvir-grazoprevir (50 mg/100 mg) — 12 week treatment of elbasvir-grazoprevir (50 mg/100 mg)
  Other Names: Zepatier

SUMMARY:
hepatitis C virus (HCV) has traditionally been treated in subspecialty health centers given the complexity of older pegylated interferon containing regimens, formerly the standard of care. This model has persisted into the modern era of direct anti-viral agents (DAAs) despite their relative simplicity, creating a bottleneck of human resources necessary to fight the largest infectious epidemic in North America. In addition, stigma and fear over cost has lead payers to restrict treatment in People Who Inject Drugs (PWIDs), even though a majority of new infections occur in this population.

This study evaluates the effectiveness of treatment of HCV with elbasvir-grasoprevir in PWIDs in a real world, community health clinic setting.

There are two prospective cohorts of PWIDs of 25 patients each, both in primary care-based community health clinics in Portland, Oregon. Cohort one is actively engaged with ambulatory medication assisted therapy with buprenorphine or extended released injectable naltrexone. Cohort two maintains active injection drug use with needle exchange and risk reduction education.

These groups are compared to a 50 patient retrospective cohort of people with substance use disorders at tertiary care hepatology-based treatment program.

All patients have genotype 1 or 4 HCV and are treated with elbasvir-grasoprevir for 12 weeks.

The investigators hypothesize there is no difference in sustained viremic response at 12 or 48 weeks post-completion of treatment (SVR 12, 48) when treating patients in a community health clinic setting as compared to the standard-of-care subspecialty setting.

DETAILED DESCRIPTION:
Hepatitis C has traditionally been treated in subspecialty health centers given the complexity of older pegylated interferon containing regimens, formerly the standard of care. This model has persisted into the modern era of direct anti-viral agents (DAAs) despite their relative simplicity, creating a bottleneck of human resources necessary to fight the largest infectious epidemic in North America. In addition, stigma and fear over cost has lead payers to restrict treatment in People Who Inject Drugs (PWIDs), even though a majority of new infections occur in this population.

This study evaluates the effectiveness of treatment of hepatitis C virus (HCV) with elbasvir-grasoprevir in people who inject drugs (PWIDs) in a real world, community health clinic setting.

There are two prospective cohorts of PWIDs of 25 patients each, both in primary care-based community health clinics in Portland, Oregon. Cohort one is actively engaged with ambulatory medication assisted therapy with buprenorphine or extended released injectable naltrexone. Cohort two maintains active injection drug use with needle exchange and risk reduction education.

These groups are compared to a 50 patient retrospective cohort of people with substance use disorders at tertiary care hepatology-based Academic Health Center.

All patients have genotype 1 or 4 HCV and are treated with elbasvir-grasoprevir for 12 weeks. The investigators exclude patients who: are under the age of 18; have a history of liver transplant; have failed past treatment of HCV; have an Aspartate aminotransferase Platelet Ratio Index (APRI) > 0.7 or APRI >0.7 but fibrosure/fibroscan of F2 or less; patients with genotype 1a and Nonstructural 5a (NS5a) resistance associated variants (RAVs); have clinical or radiologic evidence of cirrhosis; have aminotransferase levels >10x upper limit of normal; have a hemoglobin of less than 11g/dL, and are co-infected with hepatitis B or HIV.

The investigators hypothesize there is no difference in sustained viremic response at 12 or 48 weeks post-completion treatment (SVR 12, 48) when treating patients with a DAA in a community health clinic setting as compared to the standard-of-care subspecialty setting.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1b and genotype 1a without baseline NS5A resistance or Genotype 4
* APRI Score <0.7; if >0.7 a Fibrosure/Fibrotest or Fibroscan score of F2 or less
* No clinical or laboratory evidence of cirrhosis
* Readiness for treatment based on ability to make >2/3 sequential office visits
* Patients must be assessed to have decision-making capacity, be capable of consenting, and not be displaying evidence of overt intoxication.

Exclusion Criteria:

* Clinical or Laboratory Evidence of Cirrhosis
* Elevated prothrombin time unrelated to anticoagulation, hemoglobin level less than 12.3 g/L in females and <14 g/L in males, platelet count <150 × 109 cells/L), white blood cells (WBC) <4.0 x103/mm3 , aminotransferase levels more than 10 times the upper limit of normal, or albumin level <3.5 g/L.
* Previous treatment for hepatitis C infection
* Hepatocellular carcinoma
* HIV or hepatitis B virus co-infection
* Subjects taking medications that are contra-indicated to administer with Zepatier including phenytoin, carbamazepine, rifampin, St. John's Wort, and cyclosporine AND unable to change these medications to one without interactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atif Zaman, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Old Town Clinic, Portland, Oregon
  - Outside In, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
All electronic data will be maintained encrypted in the Red Cap repository. Only the primary investigator and co-investigator will have access to the master spreadsheet linking study and personal identifiers. Andrew Seaman, co-investigator and primary study contact, will be listed as the repository guardian. He will be responsible for ensuring data are released according to OHSU policy and the institutional review board (IRB) approved repository protocol, executing a repository sharing agreement in case data are released for future research, ensuring the security and confidentiality of all stored data, ensuring the security and confidentiality of data, and tracking releases of data. The repository guardian will be responsible for verifying that future releases are done in concordance with pre-proposed limits and the original consent. Data transport at the time of any future IRB approved data sharing will be approved by an updated research services agreement and separate IRB approval.

REFERENCES:
- [Background] Islam MM, Topp L, Conigrave KM, White A, Reid SE, Grummett S, Haber PS, Day CA. Linkage into specialist hepatitis C treatment services of injecting drug users attending a needle syringe program-based primary healthcare centre. J Subst Abuse Treat. 2012 Dec;43(4):440-5. doi: 10.1016/j.jsat.2012.07.007. Epub 2012 Aug 29. PMID 22938915
- [Result] Bruggmann P, Litwin AH. Models of care for the management of hepatitis C virus among people who inject drugs: one size does not fit all. Clin Infect Dis. 2013 Aug;57 Suppl 2(Suppl 2):S56-61. doi: 10.1093/cid/cit271. PMID 23884067
- [Result] Aspinall EJ, Corson S, Doyle JS, Grebely J, Hutchinson SJ, Dore GJ, Goldberg DJ, Hellard ME. Treatment of hepatitis C virus infection among people who are actively injecting drugs: a systematic review and meta-analysis. Clin Infect Dis. 2013 Aug;57 Suppl 2:S80-9. doi: 10.1093/cid/cit306. PMID 23884071
- [Result] Sylvestre DL, Litwin AH, Clements BJ, Gourevitch MN. The impact of barriers to hepatitis C virus treatment in recovering heroin users maintained on methadone. J Subst Abuse Treat. 2005 Oct;29(3):159-65. doi: 10.1016/j.jsat.2005.06.002. PMID 16183464
- [Result] Grebely J, Knight E, Genoway KA, Viljoen M, Khara M, Elliott D, Gallagher L, Storms M, Raffa JD, DeVlaming S, Duncan F, Conway B. Optimizing assessment and treatment for hepatitis C virus infection in illicit drug users: a novel model incorporating multidisciplinary care and peer support. Eur J Gastroenterol Hepatol. 2010 Mar;22(3):270-7. doi: 10.1097/meg.0b013e32832a8c4c. PMID 20425880
- [Result] Newman AI, Beckstead S, Beking D, Finch S, Knorr T, Lynch C, MacKenzie M, Mayer D, Melles B, Shore R. Treatment of chronic hepatitis C infection among current and former injection drug users within a multidisciplinary treatment model at a community health centre. Can J Gastroenterol. 2013 Apr;27(4):217-23. doi: 10.1155/2013/515636. PMID 23616960
- [Result] Mason K, Dodd Z, Sockalingam S, Altenberg J, Meaney C, Millson P, Powis J. Beyond viral response: A prospective evaluation of a community-based, multi-disciplinary, peer-driven model of HCV treatment and support. Int J Drug Policy. 2015 Oct;26(10):1007-13. doi: 10.1016/j.drugpo.2015.04.012. Epub 2015 Apr 29. PMID 26005037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for the medication assisted therapy (MAT) group were all recruited and enrolled from within a single FQHC that provides office based opioid treatment with buprenorphine. Participants in the needle exchange program were similarly recruited in that setting. Retrospective comparison group was an academic hepatology referral clinic.
Pre-assignment Details: This is a non-randomized, prospective cohort trial. No washout/run-in occured.
Period: Assessed for Eligibility --> Enrollment
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
Started | 165 | 135 | 50
Completed | 25 | 25 | 50
Not Completed | 140 | 110 | 0
Not completed — Lost to Follow-up | 17 | 36 | 0
Not completed — Inclusion Criteria: No MAT | 40 | 0 | 0
Not completed — Inclusion Criteria: neg HCV | 28 | 6 | 0
Not completed — Inclusion Criteria: No active use | 0 | 12 | 0
Not completed — Inclusion Criteria: Fibrosis > F2 | 18 | 12 | 0
Not completed — Exclusion Criteria: HIV | 4 | 4 | 0
Not completed — Inclusion Criteria: Wrong Genotype | 15 | 32 | 0
Not completed — Exclusion Criteria: NS5a Resistance | 5 | 3 | 0
Not completed — Exclusion Criteria: Treatment Readiness | 4 | 2 | 0
Not completed — Other Lab exclusion Criteria | 9 | 3 | 0
Period: Enrollment to SVR12 Results
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
Started | 25 (Pre-specified 25 participants to were enrolled.) | 25 (Pre-specified 25 participants to were enrolled.) | 50 (Prespecified 50 participants enrolled.)
Completed | 24 | 17 | 47
Not Completed | 1 | 8 | 3
Not completed — Lost to Follow-up | 1 | 8 | 3

BASELINE CHARACTERISTICS:
Population: All baseline characteristics were collected on both consented, prospective study groups (MOUD and Needle Exchange Program groups). The retrospective cohort only collected Age, Sex, Race/Ethnicity, Genotype, and APRI score and excluded level of education, duration of primary care establishment, and drug of choice.
Groups:
- Total: Total of all reporting groups
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort | Total
Number analyzed (Participants) | 25 | 25 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11.3) | 41 (11.9) | 60 (7.5) | 51 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 33 | 63
  Male | 10 | 10 | 17 | 37
Race/Ethnicity, Customized [Number; unit: participants]
  White | 22 | 22 | 50 | 84
  Black / African American | 1 | 1 | 0 | 2
  Native American | 1 | 1 | 0 | 2
  Latinx | 1 | 1 | 0 | 2
Highest Level of Education [Count of Participants; unit: Participants] — Includes 4 categories: Did not complete high school, high school completion, trade school completion, bachelors degree or higher Population: *OHSU clinic did not collect education data for comparison based on study model
  Participants
    number analyzed (Participants) | 25 | 25 | 0 | 50
    Did not complete highschool | 1 | 4 | 0 | 5
    High school completion | 18 | 11 | 0 | 29
    Trade school completion | 3 | 8 | 0 | 11
    Bachelors degree or higher | 3 | 2 | 0 | 5
Income [Count of Participants; unit: Participants] — Baseline income as percent of federal poverty level Population: *OHSU group did not collect baseline income data, as per study model
  Participants
    number analyzed (Participants) | 25 | 25 | 0 | 50
    0-50% Federal Poverty Level | 10 | 19 | 0 | 29
    51-100% Federal Poverty Level | 9 | 3 | 0 | 12
    > 101% Federal Poverty Level | 6 | 3 | 0 | 9
Fibrosis Status [Count of Participants; unit: Participants] — Baseline fibrosis predictor based on aspartate aminotransferase to platelet ratio index (APRI) below or above 0.7. All candidates had EITHER APRI < 0.7 OR non-invasive fibrosis score of F2 or below, by study inclusion data.
  Participants
    APRI < 0.7 | 19 | 23 | 30 | 72
    APRI > 0.7 | 6 | 2 | 20 | 28
Genotype [Count of Participants; unit: Participants] — Eligible participants were Genotype 1a, b, Genotype 4
  Participants
    Genotype 1a | 22 | 24 | 36 | 82
    Genotype 1b | 3 | 1 | 14 | 18
    Genotype 4 | 0 | 0 | 0 | 0
Established in Primary Care [Count of Participants; unit: Participants] — Number of participants 1) Not established in primary care, 2) established < 1 year, 3) established > 1 year. Population: *OHSU group did not collect this data per study design
  Participants
    number analyzed (Participants) | 25 | 25 | 0 | 50
    Not established in primary care | 0 | 4 | 0 | 4
    Established in primary care < 1 year | 6 | 7 | 0 | 13
    Established in primary care > 1 year | 19 | 14 | 0 | 33
Housing Status [Count of Participants; unit: Participants] — Participants were divided into either Houseless/Unstable housing (Unstable category included staying with family on short term conditional basis, couch surfing with an acquaintance, or other non-legally protected indoor housing arrangement) or Stable/Transitional housing. Population: OHSU group did not collect housing data based on our study model.
  Participants
    number analyzed (Participants) | 25 | 25 | 0 | 50
    Houseless / Unstable Housing | 4 | 8 | 0 | 12
    Transitional / Stable Housing | 21 | 17 | 0 | 38
Drug of choice [Count of Participants; unit: Participants] — Participants were asked to identify their drug of choice, given options Heroin, Methamphetamines, Alcohol, and Cannabis. Population: OHSU did not collect drug use data, as per our study model.
  Participants
    number analyzed (Participants) | 25 | 25 | 0 | 50
    Heroin | 23 | 16 | 0 | 39
    Methamphetamines | 0 | 9 | 0 | 9
    Alcohol | 1 | 0 | 0 | 1
    Cannabis | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: SVR 12
Description: Sustained Viremic Response at 12 weeks post-completion of treatment. SVR12 was determined negative if undetectable (<20 copies) by polymerase chain reaction and positive if EITHER loss-to-follow up and no lab data or virus was detected greater than 20 copies.
Time Frame: 24 weeks post-initiation of treatment (12 weeks post-completion of treatment)
Population: All participants enrolled were analyzed using intention to treat (ITT) methodology for sustained viremic response at 12 weeks after end of treatment (SVR12).
Measure: Count of Participants; unit: Participants
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
Number analyzed (Participants) | 25 | 25 | 50
Participants
  SVR12 negative, intention to treat | 24 | 15 | 47
  SVR12 positive, intention to treat | 1 | 10 | 3

2. Secondary Outcome: SVR 48
Description: Sustained Viremic Response at 48 weeks post-completion of treatment (SVR48). Participants "Achieving SVR48" had a negative hepatitis C real time polymerase chain reaction (RT-PCR) test at 48 weeks after end of treatment. Participants who "Did Not Achieve SVR48" had a positive hepatitis C RT-PCR test at 48 weeks after end of treatment.
Time Frame: 60 weeks post-initiation of treatment (48 weeks post-completion of treatment)
Population: Limitations in study funding and delayed recruitment prevented both prospective groups from collecting full SVR48 data. Therefore, PER PROTOCOL (PP) data presented below. Analysis framework for this secondary outcome was not pre-specified but PP analysis most appropriate given reasons for lacking data. OHSU comparison did not collect SVR48 data.
Measure: Count of Participants; unit: Participants
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
Number analyzed (Participants) | 17 | 7 | 0
Participants
  Achieved SVR48 | 17 | 3 | 0
  Did Not Achieve SVR48 | 0 | 4 | 0

3. Secondary Outcome: Discontinuation Rate or Lost To Follow Up
Description: Percentage of patients discontinuing medications prior to completion of 12 weeks or being lost to follow up, defined as inability to reach patient after 3 attempts and patients not following up with primary endpoint labs (SVR 12, 48)
Time Frame: Study duration (60 weeks)
Population: All participants analyzed for this variable
Measure: Count of Participants; unit: Participants
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
Number analyzed (Participants) | 25 | 25 | 50
Participants
  Completed therapy and SVR12 lab confirmation | 24 | 16 | 47
  Discontinued therapy, or incomplete SVR12 labs | 1 | 9 | 3

4. Secondary Outcome: NS5A Resistance
Description: Percentage of patients with genotype 1a and NS5A Resistance-Associated Variants (RAVs)
Time Frame: At Study Screening/Enrollment
Population: 165 potential participants in medication assisted therapy group and 135 potential participants in needle exchange group were analyzed for Non-Structural Protein 5a (NS5a) resistance. OHSU Hepatology cohort only included treated individuals and NS5a resistance data were not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
Number analyzed (Participants) | 165 | 135 | 0
Participants
  NS5a Resistance to Elbasvir-Grazoprevir Detected | 5 | 3 | 0
  NS5a Resistance to Elbasvir-Grazoprevir Absent | 160 | 132 | 0

5. Secondary Outcome: Medication Adherence
Description: Adherence determined by client/subject self-reported medication adherence measured by percentage of pills taken on a monthly basis. Categorically separated into < 90% adherence, 90-99% adherence, 100% adherence.
Time Frame: 12 weeks (duration of treatment)
Population: Enrolled study participants in prospective arms initiating therapy. Self report combined will pharmacist pill count adherence data assessed by study pharmacist at q4week study visits, including end of treatment. Retrospective comparison group at OHSU did not collect adherence data.
Measure: Count of Participants; unit: Participants
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
Number analyzed (Participants) | 25 | 25 | 0
Participants
  Less than 90% Adherence | 0 | 8 | 0
  90 - 99% adherence | 2 | 0 | 0
  100% adherence | 23 | 17 | 0

6. Secondary Outcome: Injection Drug Use Relapse (IDU)
Description: Self reported relapse IDU following HCV treatment (MAT arm)
Time Frame: Duration of study (60 weeks)
Population: These data were not collected. The study group determined that the definition of "relapse" was inappropriate for the study population given the nature of ongoing use in the MAT group and the lack of comparison with the outside in group, that was currently using drugs by definition. Scientific value of these data was thought to be limited.
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Between study enrollment and SVR12 = 24 weeks
Description: Reporting mirrors clinicaltrials.gov definitions. All-Cause Mortality and Other [Not Including Serious] Adverse Events were not monitored/assessed for the OHSU Hepatology Clinic, Academic Center Retrospective Cohort. All serious and other adverse effects were monitored for the two prospective arms, as reported below.
Arm/Group | Old Town Clinic, Medication Assisted Therapy Group | Outside In Clinic, Needle Exchange Program | OHSU Hepatology Clinic, Academic Center Retrospective Cohort
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25 | 0/0
Other Adverse Events (participants affected / at risk) | 15/25 | 18/25 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Old Town Clinic, Medication Assisted Therapy Group (N=25) | Outside In Clinic, Needle Exchange Program (N=25) | OHSU Hepatology Clinic, Academic Center Retrospective Cohort (N=0)
Infective Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — One participant developed infectious endocarditis as a complication of active injection drug use during the study period in the MAT arm.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Old Town Clinic, Medication Assisted Therapy Group (N=25) | Outside In Clinic, Needle Exchange Program (N=25) | OHSU Hepatology Clinic, Academic Center Retrospective Cohort (N=0)
Headache (Nervous system disorders) | 8 (8) | 6 (6) | 0 (0) — Mild headache, did not discontinue therapy, self-limited
Nausea (Gastrointestinal disorders) | 6 (6) | 7 (7) | 0 (0) — Mild, self limiting
Fatigue (Psychiatric disorders) | 8 (8) | 10 (10) | 0 (0) — Mild, self-limited, did not lead to discontinuation
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) — Mild, self-limited, did not lead to discontinuation
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Mild, self-limited, did not lead to discontinuation

LIMITATIONS AND CAVEATS:
Study groups comparisons of sites of enrollment/treatment (MAT clinic vs needle exchange) rather than disease state (many MAT participants used needle exchange; many needle exchange on MAT); funding limitations prevented SVR48 collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03093415/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03093415/ICF_001.pdf